CLINICAL TRIAL: NCT05712018
Title: Comparison of Different 6% Hydroxyethyl Starch (130/0.4) Coload Volumes on the 90% Effective Dose of Norepinephrine Infusion Prophylaxis for Hypotension During Spinal Anesthesia for Cesarean Section
Brief Title: Comparison of Different HES Coload Volumes on the 90% ED of Norepinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2023-1
Record Dates: First submitted 2023-01-10; First posted 2023-02-03 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Hydroxyethyl starch 130/0.4; Postspinal anesthesia hypotension; Coload; Cesarean section
MeSH Terms: interventions — Colloids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 ml/kg Hydroxyethyl starch coload group (Experimental): No fluid coload was given. An initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia
  Interventions: Drug: Hydroxyethyl starch coload - 0 ml/kg
- 5 ml/kg Hydroxyethyl starch coload group (Experimental): 5 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia.
  Interventions: Drug: Hydroxyethyl starch coload - 5 ml/kg
- 10 ml/kg Hydroxyethyl starch coload group (Experimental): 10 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia.
  Interventions: Drug: Hydroxyethyl starch coload - 10 ml/kg

INTERVENTIONS:
Drug: Hydroxyethyl starch coload - 0 ml/kg — No fluid coload was given. An initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Colloid
  Arms: 0 ml/kg Hydroxyethyl starch coload group
Drug: Hydroxyethyl starch coload - 5 ml/kg — 5 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Colloid
  Arms: 5 ml/kg Hydroxyethyl starch coload group
Drug: Hydroxyethyl starch coload - 10 ml/kg — 10 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Colloid
  Arms: 10 ml/kg Hydroxyethyl starch coload group

SUMMARY:
The purpose of this study is to investigate the effect of different 6% hydroxyethyl starch (130/0.4) coload volumes on the 90% effective dose of norepinephrine infusion prophylaxis for hypotension during spinal anesthesia for cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Coload has been highly demonstrated for prevention and/or treatment of post-spinal anesthesia hypotension. In addition, there's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. The purpose of this study is to investigate the effect of different 6% hydroxyethyl starch (130/0.4) coload volumes on the 90% effective dose of norepinephrine infusion prophylaxis for hypotension during spinal anesthesia for cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥180 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
ED 50 | 1-15 minutes after spinal anesthesia
  The dose of prophylactic norepinephrine that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) of patients
ED 90 | 1-15 minutes after spinal anesthesia
  The dose of prophylactic norepinephrine that would be effective in preventing postspinal anesthesia hypotension in 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min
The incidence of nausea and vomiting | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline
pH | Immediately after delivery
  From umbilical arterial blood gases
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University; Xiangsheng Xiong, M.D., Study Chair — The Fifth People's Hospital of Huaian
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China